CLINICAL TRIAL: NCT00763841
Title: A Pilot Study Using Transcranial Magnetic Stimulation (TMS) to Investigate the Role of the Temporal Cortex in Schizophrenic Patients With Auditory Hallucinations
Brief Title: Transcranial Magnetic Stimulation (TMS) for Treatment of Auditory Hallucinations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: NSW Schizophrenia Fellowship (Unknown); Rebecca Cooper Medical Research Foundation (Unknown)
Responsible Party: Assoc. Prof. Colleen Loo, University of NSW
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07019
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-11

CONDITIONS: Auditory Hallucinations
Keywords: Auditory hallucinations
MeSH Terms: conditions — Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stimulation will be given daily at a particular site for three days a week
  Interventions: Device: Transcranial magnetic stimulation
- 2 (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Stimulation will be given daily at a particular site for three days a week
  Arms: 1
Device: Sham
  Arms: 2

SUMMARY:
Transcranial magnetic stimulation (TMS) involves the use of magnetic fields to non-invasively stimulate the brain. Studies overseas have suggested this may be an effective and safe treatment for auditory hallucinations in patients with schizophrenia. This is a sham-controlled, double-blind trial of TMS stimulation for the treatment of auditory hallucinations in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Over 18, with DSM-IV diagnosis of Schizophrenia and auditory hallucinations of clear external origins, refractory to pharmacotherapy and occurring at least 5 times per day.

Exclusion Criteria:

* Subjects with contraindications to TMS (e.g. epilepsy, pacemaker) or those with an unacceptably high risk (e.g. suicide risk) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 1999-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Daily Voices Ratings (Mental Health Research Institute, Victoria) | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MBBS, FRANZCP. MD, Principal Investigator — University of NSW
Locations (1):
- School of Psychiatry, Sydney, New South Wales, Australia